CLINICAL TRIAL: NCT02370446
Title: Testing a Personalize Medication Log for Patients With Lymphoma
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-008
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Lymphoma
Keywords: Medication Log; 15-008
MeSH Terms: conditions — Lymphoma | interventions — Standard of Care; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- patient gets personalized medication log: Patients in the intervention group will receive a personalized medication log that includes all treatment medications (IV and oral), days of treatment and medication specific information such as timing or diet restrictions. The personalized medication log and patient education materials (fact cards) will be placed in a clear plastic envelope that the patient can carry with them throughout treatment.
  Interventions: Other: personalized medication log; Behavioral: questionnaires; Behavioral: Cognitive Interview
- patient gets standard of care: Current MSKCC standards of professional nursing practice require the professional nurse to develop a plan of care that includes teaching the patient and support system the prescribed prescriptions / regimen and all doses, route, length of treatment, side effects and safety precautions.
  Interventions: Other: standard of care; Behavioral: questionnaires

INTERVENTIONS:
Other: personalized medication log
  Groups: patient gets personalized medication log
Other: standard of care
  Groups: patient gets standard of care
Behavioral: questionnaires
Behavioral: Cognitive Interview
  Groups: patient gets personalized medication log

SUMMARY:
The purpose of this study is to see if using the MedLog is helpful to patients. Since the investigators do not yet know if this MedLog is helpful, some patients will receive it and some will receive our standard of care. The investigators want to know whether providing patients with this additional information is helpful and if having this additional information about their treatment schedule has an effect on their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lymphoma
* No prior treatment for lymphoma
* Scheduled to receive CHOP14 +/- Rituximab, CEOP 21, CHOPE or EPOCH +/- Rituximab
* Age 18 or older
* Able to speak and read English

Exclusion Criteria:

* Documented major psychopathology or cognitive impairment likely in the judgment of the research staff to interfere with the participation or completion of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan-Kettering Cancer Center (MSKCC).
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
patient satisfaction with medication log ( identified qualitatively through the process of cognitive interviewing and further measured with the satisfaction question on the Patient Satisfaction and Treatment Data Sheet) | 1 year
  as identified qualitatively through the process of cognitive interviewing and further measured with the satisfaction question on the Patient Satisfaction and Treatment Data Sheet

SECONDARY OUTCOMES:
changes in quality of life | 1 year
  before and during therapy, as measured by PROMIS, Distress Thermometer and FACT scores, and to evaluate adherence with oral treatment medications, as measured by the MMAS-8.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Anselmi, RN, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/